CLINICAL TRIAL: NCT05044260
Title: Evaluation of Direct Sinus Lift Using Ptfe Titanium Reinfored Membrane Assosiated With Immediate Implant Placement (Clinical Trial)
Brief Title: Sinus Lift Using PTFE Titanium Reinforced Membrane
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: sinus_lift2020
Record Dates: First submitted 2021-09-06; First posted 2021-09-14 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Sinus Lift

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Direct Sinus elevation using SLA Kit (Experimental)
  Interventions: Procedure: Direct sinus lift with titanium reinforced PTFE membrane

INTERVENTIONS:
Procedure: Direct sinus lift with titanium reinforced PTFE membrane — Implants will be placed immediately after sinus lifting procedure and maintaining the sinus membrane in position using PTFE titanium reinforced membrane.

SUMMARY:
Various attempts have been implemented using different materials and techniques to augment the maxillary sinus floor enhancing autogenous bone formation to allow proper dental implant positioning. The aim of this study is to evaluate the sinus lift procedure using polytetrafluoroethylene (PTFE) titanium-reinforced membrane to maintain the space formed after Schneiderian membrane elevation followed by immediate implant placement.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders requiring implant placement in posterior maxilla
* Age range: 40-60 years.
* Good oral hygiene
* Healthy maxillary sinus free from pathology
* The minimum crestal bone height is (4-6) mm
* Patients who are willing and fully capable to comply with the study protocol.

Exclusion Criteria:

* Sinus infection
* Tumors or pathologic lesions in sinus
* Severe allergic rhinitis.
* Chronic topical steroid use.
* Radiation therapy.
* Psychologic / mental impairment
* Acute infection (periodontitis or mucosal infection
* Patients on radiotherapy or chemotherapy.
* Alcohol or drug abuse.
* Patient with systemic disorder (uncontrolled Diabetes mellitus, autoimmune diseases, bone diseases, etc.)
* Smokers
* Parafuctional habits

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-10-20 (Estimated); Study Completion 2021-10-20 (Estimated)

PRIMARY OUTCOMES:
Change in implant stability | at baseline and 6 months
  It will be measured using Osstell
Change in bone formation | at baseline and 6 months
  It will be measured uisng CBCT on Demand 3d software
Change in bone height | at baseline and 6 months
  It will be measured uisng CBCT on Demand 3d software
Change in bone density | at baseline and 6 months
  It will be measured uisng CBCT on Demand 3d software

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt